CLINICAL TRIAL: NCT01029483
Title: Energy and Appetite Regulation by Low CHO Diets
Brief Title: The Energy Balance Study
Acronym: EBS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Diane D. Stadler, OHSU
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT002753 (NIH)
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2009-12-10 (Estimated); Status verified 2009-12

CONDITIONS: Obesity
Keywords: Obesity; Weight loss; low carbohydrate diets; high complex carbohydrate diets; Healthy adults; Body composition; Energy Expenditure
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Diet, Carbohydrate-Restricted; Diet, High-Protein Low-Carbohydrate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low carbohydrate diet (Experimental): 6 week ad libitum low carbohydrate diet; research diet provided at 120% of estimated energy requirement for weight maintenance; carbohydrate intake limited to 28g/d
  Interventions: Other: Low carbohydrate diet
- High Carbohydrate Diet-ad libitum (Active Comparator): High complex carbohydrate diet (55% carbohydrate, 18% protein, 27% fat. 120% of estimated energy needs for weight maintenance provided, participants allowed to eat as much or as little as desired to satisfy appetite
  Interventions: Other: High-carbohydrate ad libitum intervention
- High Carbohydrate Diet-Energy-matched (Active Comparator): High carbohydrate diet (55% carbohydrate, 18% protein and 27% fat). Energy intake restricted to ~68% of energy needs for weight maintenance. Participants required to eat all food provided and nothing else
  Interventions: Other: High carbohydrate diet-energy matched intervention

INTERVENTIONS:
Other: Low carbohydrate diet — Ad libitum low carbohydrate diet (<28g carbohydrate/day). Participants provided with research diet at 120% of estimated energy needs for weight maintenance and allowed to eat as much or as little of the food desired.
  Other Names: Low CHO diet; Atkins Diet
  Arms: Low carbohydrate diet
Other: High-carbohydrate ad libitum intervention — Participants provided with a high complex carbohydrate diet (55% carbohydrate, 18% protein, and 27% fat) at 120% of estimated energy needs for weight maintenance and allowed to eat as much or as little of the foods provided as desired
  Other Names: High CHO-ad lib diet; DASH-ad lib diet
  Arms: High Carbohydrate Diet-ad libitum
Other: High carbohydrate diet-energy matched intervention — Participants provided a high complex carbohydrate diet (55% carbohydrate, 18% protein, and 27% fat) at ~70% of estimated energy needs to maintain weight. Participants required to eat all food provided and nothing else.
  Other Names: High CHO energy-matched diet; DASH energy-mathched diet
  Arms: High Carbohydrate Diet-Energy-matched

SUMMARY:
Very low carbohydrate diets and high-complex carbohydrate, low-fat diets are popular weight-loss methods in the United States. The purpose of the Energy Balance Study is to explore how extreme differences in diet affect eating behaviors, activity and calorie-use, and body composition.

We will conduct a controlled feeding study (all food will be provided for the duration of the study) in which obese adults will be randomly assigned to one of three dietary groups: a low-carbohydrate-eat as much as you like diet, a high-carbohydrate-eat as much as you like diet, or a high-carbohydrate-calorie-restricted diet. The low-carbohydrate diet will be modeled after the Induction Phase of the Atkins Diet. The high carbohydrate diet will be based on the "Dietary Approaches to Stop Hypertension (DASH)" diet. During the first 3 weeks, participants will eat a typical diet adjusted so that they neither gain or lose weight. Then, for 6 weeks, they will eat their assigned research diet. Resting calorie use and body composition measurements will be taken at the end of week 2 and week 9. Frequent blood sampling for 24 hours will be done through a catheter (tube) placed in an arm vein at the end of weeks 2 and week 9 and for 12 hours at the end of week 3.

Change in body composition, activity and energy expenditure, and blood components known to influence eating behavior will be measured under typical diet conditions and after one-day and 6 weeks of the research diet.

ELIGIBILITY:
Inclusion Criteria:

* BMI; 30-50 kg/m2
* Age at least 21 years
* Relative good health

Exclusion Criteria:

* Major debilitating mental or physical illness that would interfere with participation
* Renal or hepatic disease, diabetes
* History of gallbladder disease/removal
* Hyper-or hypothyroidism
* Poorly controlled hypertension
* Use of lipid lowering medications
* Pregnancy or lactation
* Current excessive use of alcohol
* Current/recent chronic use of tobacco

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
weightloss | 6 weeks

SECONDARY OUTCOMES:
weight regulation hormones (insulin, leptin, ghrelin, GLP-1, PYY) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diane D Stadler, PhD, Principal Investigator — Oregon Health and Science University